CLINICAL TRIAL: NCT03933969
Title: Functional Predictive Value of Collective Outcome Measure(s) Status Post Total Hip/Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ryan C. McCoy, Principal Investigator, Mayo Clinic
Other Study IDs: 18-009437
Record Dates: First submitted 2019-04-30; First posted 2019-05-01 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Joint Arthroplasty; Knee and Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Researchers are trying to assess a predictive value or correlation of outcome measures results on subjects following a total knee or total hip arthroplasty in order to better predict the time frame taken to achieve certain functional milestones that are pertinent to subject population.

DETAILED DESCRIPTION:
Subjects will undergo testing for a normal physical therapy clinical assessment that is standard of care for anyone who has a total hip or total knee surgery. Researchers will be using the data obtained from standard therapy care and see if correlations exist from that data and the time taken to complete specific functional tasks.

ELIGIBILITY:
Inclusion Criteria:

* Patient's 18 years or older
* Patients who recently underwent a primary total hip or total knee arthroplasty
* Patient who recently underwent a total hip or total knee revision

Exclusion Criteria:

* Patients who lack the ability to provide informed consent
* Patients with previous total joint replacement within the last 6 months
* Patients with complications following surgery such as DVT/PE/Infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects status post total hip and total knee arthroplasty that will undergo standard inpatient and outpatient physical therapy evaluation following total joint surgery.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Assistive Device Weaning | Approximately 3 months
  Number of days to weaning from all assistive devices

SECONDARY OUTCOMES:
Weaning from pain medication, ability to reciprocally use steps, ability to walk 1 mile or 30 minutes consecutively | Approximately 3-6 months
  Number of days taken to achieve milestones

CONTACTS AND LOCATIONS:
Overall Officials: Ryan C McCoy, PT, DPT, OCS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials